CLINICAL TRIAL: NCT03026075
Title: Evaluation of the Performance of the Motus Cleansing System
Brief Title: Evaluation of the Performance of the Motus Cleansing System (MCS)
Acronym: MCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Motus GI Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CL00016
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2017-06

CONDITIONS: CRC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Colonoscopy with MCS (Experimental): Standard colonoscopy procedure with Motus Cleansing System
  Interventions: Device: Motus Cleansing System (MCS)

INTERVENTIONS:
Device: Motus Cleansing System (MCS) — The MCS enables colon cleansing during standard colonoscopy using a standard colonoscope. The cleansing device, which is attached to the tip of the colonoscope and is connected to an external workstation, generates fluid jets within the colon thus dissolving the feces into small parts. The fecal matter & fluids are drained through the evacuation pipe of the cleansing device into a collecting reservoir.

SUMMARY:
The study is multi-center study ,planned as a single arm, open trial, aimed at evaluating the performance and safety of a colon cleansing device during a colonoscopy procedure in a poorly prepared colons.

DETAILED DESCRIPTION:
Total of 47 subjects are planned to be enrolled at 3 clinical sites (1 in Germany and 2 in the Netherlands).

Subjects who meet the eligibility criteria will be screened for study participation at a baseline visit(visit 1). Subject who is eligible to the study will required to follow a specific reduced preparation instruction starting 2 days prior to the colonoscopy with the Motus Cleansing System (MCS) procedure.

Following the procedure a telephone follow-up will be conducted at 48 hours (± 24 hours) and 14 days (± 3 days) post MCS procedure to assess patient well-being and capture any Adverse Events (AE).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects being considered for diagnostic, screening or surveillance colonoscopy
2. Subjects in the age range of 18-75 years inclusive
3. Subjects with BodyMass Index (BMI) within the range of 18.5-35 inclusive
4. Subject has signed the informed consent

Exclusion Criteria:

1. Subjects with known Inflammatory Bowel Disease
2. Subjects with known diverticulitis disease or with prior incomplete colonoscopy due to diverticular disease
3. Subjects with known or detected (during colonoscopy) bowel obstruction
4. History of prior surgery to colon and/or rectum
5. ASA≥IV
6. Renal insufficiency (Creatinine ≥ 1.5mg /dL) (based on medical history)
7. Abnormal Liver enzymes (ALT/AST ≥ 2 times upper limits of normal) (based on medical history)
8. Subjects taking anticoagulants drugs (excluding aspirin) or dual antiplatelet therapy
9. Subjects with known coagulation disorder (INR >1.5).
10. Subjects treated with H2 receptor antagonists or proton pump inhibitors within the 72 hours prior to consuming the Bisacodyl
11. Subjects with active, ongoing lower GI bleeding with hemodynamic instability.
12. Subjects with known Mega Colon
13. Pregnancy (as stated by patient) or breast feeding
14. Subjects with altered mental status/inability to provide informed consent
15. Patients who have participated in another interventional clinical study in the last 2 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravit Peled, Study Director — Motus GI Technologies Ltd.
Locations (3):
- UMC Of JOHANNES GUTENBERG-UNIVERSITY MAINZ, Mainz, Germany
- Netherlands (2):
  - University Medical Centre (UMC) Radboud Department of Gastroenterology and Hepatology, Nijmegen
  - Erasmus medical center, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Keulen KE, Neumann H, Schattenberg JM, van Esch AAJ, Kievit W, Spaander MCW, Siersema PD. A novel device for intracolonoscopy cleansing of inadequately prepared colonoscopy patients: a feasibility study. Endoscopy. 2019 Jan;51(1):85-92. doi: 10.1055/a-0632-1927. Epub 2018 Jul 11. PMID 29996152

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients indicated for screening/ surveillance or diagnosis colonoscopy enrolled at 3 clinical sites as follows:
  * Radboud University Medical Center(UMC)- Netherlands-16 cases
  * Erasmus Medical Center (MC)-Netherlands-16 cases
  * Mainz University Medical Center(UMC)-Germany- 15 cases
  enrollment period : 20 December 2016 - 31 May 2017
Pre-assignment Details: The patients had reduced preparation in order to mimic poor bowel cleansing. the study bowel preparation consisted of dietary restrictions (no dried fruit, seeds or nuts) starting 2 days prior to colonoscopy, a 24-hour clear liquid diet and a split dose of 20 mg Bisacodyl (10 mg in each dose).
Period: Overall Study
Arm/Group | Colonoscopy With MCS
Started | 47
Completed | 46
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Colonoscopy With MCS
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White Non-Hispanic | 44
  Ethnicity: Hispanic | 2
  Ethnicity: Asian | 1
Region of Enrollment [Number; unit: participants]
  Netherlands | 32
  Germany | 15
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.0 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Performance of MCS in Cleansing a Poorly Prepared Colon.
Description: The rate of adequate cleansing level per subject will be evaluated by the Boston Bowel Preparation (BBPS) scoring index before and post the cleansing operation.
Time Frame: Up to 2 hours
Population: the bowel preparation level before and after the use of Motus Cleansing System was evaluated using the Boston Bowel Preparation Scale (BBPS) where patients consider to have adequate cleansing level if all 3 colon segments graded 2 or 3 ( good or excellent)
Measure: Count of Participants; unit: Participants
Arm/Group | Colonoscopy With MCS
Number analyzed (Participants) | 46
Participants
  adequate cleaning after the use of MCS | 46
  adequate cleaning at baseline | 9
Statistical Analysis 1: Comparison: Colonoscopy With MCS; The primary objective of the study is to evaluate the effectiveness of MCS in cleansing a poorly prepared colon. A sample size of 47 patients is required as per a McNemar test to determine that the paired discordant proportions are significantly different under the followings assumptions: Probability of Type I Error (α) = 0.05, Power (1 - β) = 0.8 Proportion switching from + to - = 0, Proportion switching from - to + = 0.6 Potential of dropout 10% (i.e. 4 cases); Test type: Superiority; p < 0.01, McNemar

ADVERSE EVENTS:
Time Frame: Follow up was conducted immediately after the procedure before patient discharge and at 2-3 days and 14-16 days post procedure
Arm/Group | Colonoscopy With MCS
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 5/47
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colonoscopy With MCS (N=47)
Bloating (Gastrointestinal disorders) | 5 (5) — abdominal discomfort and or stomach discomfort

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT03026075/Prot_SAP_000.pdf